CLINICAL TRIAL: NCT05893784
Title: The Effect of Progressive Relaxation Exercises Applied to Individuals With Diabetes on Fatigue and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bahar İNKAYA, Doç.Dr, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AnkaraYBU1324356
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; nurse; progressive relaxation exercises; fatigue; sleep
MeSH Terms: conditions — Diabetes Mellitus; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- END (Experimental): Use of progressive relaxation exercises education
  Interventions: Other: Use of progressive relaxation exercises education
- END free (No Intervention): patient witout of progressive relaxation exercises education

INTERVENTIONS:
Other: Use of progressive relaxation exercises education — Progressive relaxation exercises education It starts with deep breathing exercises along with music. Then stretching and relaxation exercises are performed. After the education, an 8-minute video in which the progressive relaxation exercises was explained practically to the individuals was sent to their mobile phones. The participants were asked to perform these exercises regularly for 4 weeks, each day one hour before going to bed, simultaneously with the video.
  Arms: END

SUMMARY:
The aim of this study was to examine the effect of the progressive relaxation exercises applied to the individuals with diabetes on fatigue and sleep. This randomized controlled study was a single-blind, parallel intervention and control group experimental study. The researcher applied the training for the progressive relaxation exercises to the intervention group. Socio-demographic data, 'Pittsburgh Sleep Quality Index' and 'The Fatigue Severity Scale' were used for the study.

DETAILED DESCRIPTION:
The study was conducted on patients who applied to the endocrine polyclinic of a hospital in Turkey and voluntarily agreed to participate in the study. The patients were diagnosed with type 1 or type 2 diabetes, were over 18 years old and were using insulin. The patients were able to communicate and had no disease that could prevent them from exercising.

The Intervention (n=33) and control groups (n=30) were formed by simple randomization method.

Data was collected by using "Patient Identification Form", "Pittsburgh Sleep Quality Index" and "The Fatigue Severity Scale".

Patient Identification Form was created by scanning the literature for this study. In this form, there were 10 questions in total. The questions included the first letters of the name and surname of the patient for coding purposes. The other questions were about age, marital status, employment status, educational status, drinking and smoking habbits, participation in exercise training, exercise and sleep patterns.

Pittsburgh Sleep Quality Index was developed by Buysse et al. in 1989. It was adapted into Turkish by Ağargün et al. in 1996 as PUKI. PUKI was a 24-item scale and it was used to evaluate sleep quality and disturbance of the previous month. 19 of the questions were self-report questions and those were answered by the patient. The question number 19 was about the availability of a roommate or spouse and it was not used in scoring. The remaining 5 questions of 24 were to be answered by a spouse or a roommate, they were also not included in the scoring. The 18 scored questions of the scale consisted of 7 components which were Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component was evaluated with a score between 0 and 3 points. The total score of the 7 components was accepted as the score of the scale. Therefore the total score of the scale was between 0 and 21 points. A total score greater than 5 was accepted to be "poor sleep quality". The Cronbach Alpha internal consistency coefficient of the scale was found to be 0.80.

Fatigue Severity Scale was developed by Krupp in 1989. It was adapted into Turkish by Armutlu et al. in 2007. The Fatigue Severity Scale was cited as the best example among one-dimensional scales. This scale consisted of 9 questions in total and the person indicated how much he or she agreed with each question by choosing a value between 1 and 7 where 1 means I totally disagreed and 7 means I totally agreed. The score range of the scale was between 9 and 63 points. A score of 36 or higher indicated severe fatigue. The total score was calculated by taking the average of 9 answers. The cut-off value for pathological fatigue was determined as 4 and above. The lower the total score, the less fatigue. Cronbach's alpha reliability coefficient of the SSS is 0.96.

Progressive relaxation exercises training and questionnaires were administered to the experimental group face-to-face in the endocrine polyclinic examination room by the researcher, and each interview lasted approximately 30 minutes.

Written consent was obtained from the participants before the research. After explaining the benefits, application steps, frequency and duration of progressive relaxation exercises, practical exercise training was given by the researcher.

After the training, an 8-minute video in which the progressive relaxation exercises was explained practically to the individuals was sent to their mobile phones. The participants were asked to perform these exercises regularly for 4 weeks, each day one hour before going to bed, simultaneously with the video.

The aforementioned video included breathing exercises and progressive muscle stretching exercises, with music in the background to relax the patient. After 4 weeks, when the individuals in the experimental group came to the endocrine polyclinic for control, Pittsburgh Sleep Quality Index and The Fatigue Severity Scale were applied again by the researcher as a post-test. No training was given to the control group by the researcher during the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 or type 2 diabetes
* using insulin
* had no disease that could prevent them from exercising.

Exclusion Criteria:

* Not having been diagnosed with diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | a day before the education
  Patient Identification Form was created by scanning the literature for this study. In this form, there were 10 questions in total. The questions included the first letters of the name and surname of the patient for coding purposes. The other questions were about age, marital status, employment status, educational status, drinking and smoking habbits, participation in exercise training, exercise and sleep patterns.
Pittsburgh Sleep Quality Index | a day before the education
  Pittsburgh Sleep Quality Index was a 24-item scale and it was used to evaluate sleep quality and disturbance of the previous month. 19 of the questions were self-report questions and those were answered by the patient. The question number 19 was about the availability of a roommate or spouse and it was not used in scoring. The remaining 5 questions of 24 were to be answered by a spouse or a roommate, they were also not included in the scoring. The 18 scored questions of the scale consisted of 7 components which were Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component was evaluated with a score between 0 and 3 points. The total score of the 7 components was accepted as the score of the scale. Therefore the total score of the scale was between 0 and 21 points. A total score greater than 5 was accepted to be "poor sleep quality".
Fatigue Severity Scale | a day before the education
  Fatigue Severity Scale was cited as the best example among one-dimensional scales. This scale consisted of 9 questions in total and the person indicated how much he or she agreed with each question by choosing a value between 1 and 7 where 1 means I totally disagreed and 7 means I totally agreed. The score range of the scale was between 9 and 63 points. A score of 36 or higher indicated severe fatigue. The total score was calculated by taking the average of 9 answers. The cut-off value for pathological fatigue was determined as 4 and above.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No